CLINICAL TRIAL: NCT07295964
Title: Influence of AI Driven Software Programs and Digital Occlusal Collision Corrections on the Occlusal Adjustment of 3D-Printed Restorations: A Clinical Trial
Brief Title: Accuracy of Intraoral Scan Post-processing Methods: A Clinical Trial
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: National and Kapodistrian University of Athens (Other)
Responsible Party: Principal Investigator, Panagiotis Ntovas, PhD Canditate, Department of Operative Dentistry, School of Dentistry, Greece, National and Kapodistrian University of Athens
Allocation: Randomized | Model: Single Group | Masking: Quadruple | Purpose: Treatment
Other Study IDs: STUDY3534
Record Dates: First submitted 2025-01-09; First posted 2025-12-22 (Actual); Last update posted 2025-12-22 (Actual); Status verified 2025-12

CONDITIONS: Restoration Design; Digital Occlusal Collision
Keywords: Artificial intelligence; Prosthodontics; Automated Design; Occlusion Collusion

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- AI driven design (Experimental): The restoration is designed using an AI driven software
  Interventions: Other: Artificial intelligence driven registration
- AI driven refinement of maxillomandibular relatioship (Experimental): The restoration is design using a maxillomandibular relationship refined by an AI tool
  Interventions: Other: Artificial intelligence driven registration
- Design of a restoration after automated collision correction (Experimental): The restoration is designed using the maxillomandibular relationship obtained after the use of a software for automated collision correction
  Interventions: Other: Software based registration
- Design of a restoration using the registration without any further refinement (Active Comparator): The restoration is designed using the conventional maxillomandibular relationship as it i obtained by the intraoral scanning without further refinement
  Interventions: Other: Software based registration

INTERVENTIONS:
Other: Artificial intelligence driven registration — Maxillomandibular relationship is refined using AI driven tools
  Arms: AI driven design; AI driven refinement of maxillomandibular relatioship
Other: Software based registration — Maxillomandibular relationship is refined using software based algorithms
  Arms: Design of a restoration after automated collision correction; Design of a restoration using the registration without any further refinement

SUMMARY:
In the last decade, progressive developments in computer hardware, software, manufacturing technologies, and dental materials consistently enhanced the use of digital technologies in dentistry. Traditional prosthodontic techniques have relied on manual fabrication processes, which often resulted in challenges such as suboptimal prosthesis fit, compromised occlusal stability, and limited customization options. However, the advent of 3D printing technology has revolutionized the field, offering new possibilities for patient-specific prosthodontic rehabilitation.

An accurate maxillomandibular relationship between the maxillary and mandibular casts is fundamental to prosthodontic practice. In the integration of intraoral scanners (IOSs) for different dental interventions, the accuracy of the digitizing methods recording the maxillomandibular relationship is similarly essential. The maxillomandibular relationship accuracy recorded by using IOSs has been analyzed in various in vitro and clinical studies.

Intraoral digital scans are recorded in an unload condition, with the mouth open, while acquiring the maxillary and the mandibular intraoral scans. This condition changes when capturing the virtual occlusal records at maximum intercuspation position (MIP). Occlusal collisions are caused by the tooth location discrepancy resulting from the periodontal ligament plasticity between the recording of the intraoral digital scans and the virtual occlusal records, as well as from the intraoral scanning distortion and alignment procedures.

Artificial intelligence driven program software and occlusal collisions or mesh interpenetrations tools have been proposed to improve the maxillomandibular relationship of the scanned models. The software programs of the IOSs can automatically eliminate the occlusal collisions present in virtual articulated casts. Similarly, dental computer-aided design (CAD) programs can automatically detect and eliminate occlusal collisions among the articulated intraoral digital scans imported. However, the effect of the occlusal collision corrections performed by using IOSs or CAD programs on the occlusal adjustment of the restorations is unknown.

DETAILED DESCRIPTION:
Objectives The goal of this clinical investigation is to assess the impact of occlusal collision corrections performed by the software program of 2 intraoral scanners (TRIOS 4; 3Shape A/S, i700; Medit) and two dental CAD programs (DentalCAD, Rijeka; exocad & Dental System ;3Shape), for maxillomandibular relationship acquired at maximum intercuspation position, on the intraoral occlusal adjustment of 3D-printed restorations. The null hypothesis was that no difference would be found for the intraoral occlusal adjustment of the assessed 3D-printed restorations, designed by the different collision correction methods, independently of the IOS and the dental CAD software.

Materials and methods In total 30 patients are going to be enrolled in the present study. Initially, two intraoral scanners will be used to record the experimental digital scans: TRIOS 4 (TRIOS 4, wireless, v. 22.2.3; 3Shape A/S) and i700 (i700, Medit). Two groups will be established depending on the correction of the occlusal collisions performed by using the IOS software program: not corrected and corrected group. Moreover, 3 subgroups will be established based on the following correction procedures performed in a dental CAD program (DentalCAD, Rijeka; exocad GmbH): no changes, cast trimming (trimming subgroup), opening of the vertical dimension (opening subgroup).

For each record a model-free complete digital workflow will be employed to print a crown using a 3D printer (Pro 2, Sprintray) with a compatible resin (KeyDenture Try-in, KeystoneIndustries). Each restoration is going to be tried and fit intraorally. The sequence of try-in will be randomized. Initially, after adjusting for distal and mesial approximal contact areas, the internal fit will be checked and adjusted to eliminate any interferences in order to ensure the optimal fitting of the restorations. After ensuring optimal fitting, the investigator will take an intraoral quadrant scan including the crown.

The occlusal adjustment strategy will be as follows: Under normal occlusal forces, 8 μm articulating film (AccuFilm, FastCheck, Parkell) will be used consecutively, followed by occlusal contact check using 8 μm articulation foil (Shimstock-foil, Bausch, Cologne, Germany) under strong occlusal forces. Then the occlusal adjustments will be made with fine diamond burs and will polished. After that, the same investigator will take in intraoral digital quadrant scan to record the post-adjustment volume of the each crown.

For the qualitative analysis, color-coded maps of the superimposed pre- and post-adjustment .STL files will be used, utilizing metrology software (Geomagic, 3DSystems). The primary outcome measure will be the volumetric measurement (mm3) of occlusal adjustment amount of the tested 3D printed restorations. The color codes will be standardized in every evaluation, and the occlusal views of color-coded maps will be evaluated by two investigators independently. Less than 0.3 mm differences which were presented in green and yellow, are going to be considered clinically as irrelevant. Meanwhile, turquoise (0.3-04mm), dark blue (0.4-0.5 mm), and red (>0.5 mm) will be taken into consideration for the evaluation. The investigators will rate the adjustment amount 0-4 scores based on the adjustment surface, and the geometrical characteristics of the adjustment. Grade 4 adjustments will be considered to require renewal of the restoration due to a change in the anatomical contour of the reconstructions, whereas Grade 0 will be considered as perfect.

Inclusion criteria Age > 18 years old Absence of painful temporomandibular disorder Presence of natural opposing teeth Presence of a stable maximum intercuspation relationship Exclusion criteria Pain in orofacial region Visible periapical lesion < Class II mobility

Statistical Analysis The descriptive statistics will be given as mean (standard deviation) and median [first and third quartiles] for continuous variables, while frequency and percentages will be given for categorical variables. The 2 × 2 cross-table variance analyses and Greenhouse Geisser corrections will be tested for the carry-over effect. The two dependent and independent variables will be compared via the Wilcoxon and Mann-Whitney U tests, respectively. For the 2 × 2 crossover design, repeated measure ANOVA will be implemented. The Wilcoxon test analyzed the operator and patient preferences outcomes. Statistical analysis will be performed using a statistical software program (SPSS Statistics, v23.0; IBM Corp, New York, USA). The significance level will set at p<0.05.

ELIGIBILITY:
Inclusion Criteria:

Age > 18 years old Absence of painful temporomandibular disorder Presence of opposing teeth Presence of a stable maximum intercuspation relationship

Exclusion Criteria:

- Pain in orofacial region Visible periapical lesion < Class II mobility

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2026-01-25 (Estimated); Primary Completion 2026-12-25 (Estimated); Study Completion 2027-06-25 (Estimated)

PRIMARY OUTCOMES:
Level of adjustment | Baseline, after the adjustment of the try-in restorations
  The investigators will rate the adjustment amount 0-4 scores based on the adjustment surface, and the geometrical characteristics of the adjustment. Grade 4 adjustments will be considered to require renewal of the restoration due to a change in the anatomical contour of the reconstructions, whereas Grade 0 will be considered as perfect.

CONTACTS AND LOCATIONS:
Locations (1):
- Clinic, Athens, Attica, Greece

IPD SHARING:
Plan to Share IPD: Yes
Only IPD used in the results publication
Supporting Information: Study Protocol, ICF, CSR

REFERENCES:
- [Background] Yuzbasioglu E, Kurt H, Turunc R, Bilir H. Comparison of digital and conventional impression techniques: evaluation of patients' perception, treatment comfort, effectiveness and clinical outcomes. BMC Oral Health. 2014 Jan 30;14:10. doi: 10.1186/1472-6831-14-10. PMID 24479892
- [Background] Sakrana AA. In vitro evaluation of the marginal and internal discrepancies of different esthetic restorations. J Appl Oral Sci. 2013 Nov-Dec;21(6):575-80. doi: 10.1590/1679-775720130064. PMID 24473725
- [Background] Kokubo Y, Ohkubo C, Tsumita M, Miyashita A, Vult von Steyern P, Fukushima S. Clinical marginal and internal gaps of Procera AllCeram crowns. J Oral Rehabil. 2005 Jul;32(7):526-30. doi: 10.1111/j.1365-2842.2005.01458.x. PMID 15975133
- [Background] Mai HN, Lee KB, Lee DH. Fit of interim crowns fabricated using photopolymer-jetting 3D printing. J Prosthet Dent. 2017 Aug;118(2):208-215. doi: 10.1016/j.prosdent.2016.10.030. Epub 2017 Jan 12. PMID 28089333
- [Background] van Noort R. The future of dental devices is digital. Dent Mater. 2012 Jan;28(1):3-12. doi: 10.1016/j.dental.2011.10.014. Epub 2011 Nov 26. PMID 22119539
- [Background] Ng J, Ruse D, Wyatt C. A comparison of the marginal fit of crowns fabricated with digital and conventional methods. J Prosthet Dent. 2014 Sep;112(3):555-60. doi: 10.1016/j.prosdent.2013.12.002. Epub 2014 Mar 11. PMID 24630399
- [Background] Delong R, Ko CC, Anderson GC, Hodges JS, Douglas WH. Comparing maximum intercuspal contacts of virtual dental patients and mounted dental casts. J Prosthet Dent. 2002 Dec;88(6):622-30. doi: 10.1067/mpr.2002.129379. PMID 12488856
- [Background] van den Bergh HT, Owen CP, Howes DG. A comparison of different methods and materials for establishing maximal intercuspal position: A clinical study. J Prosthet Dent. 2024 Oct;132(4):749-754. doi: 10.1016/j.prosdent.2022.01.036. Epub 2022 Sep 30. PMID 36184310
- [Background] Morsy N, El Kateb M. Accuracy of intraoral scanners for static virtual articulation: A systematic review and meta-analysis of multiple outcomes. J Prosthet Dent. 2024 Sep;132(3):546-552. doi: 10.1016/j.prosdent.2022.09.005. Epub 2022 Nov 2. PMID 36333175
- [Background] Revilla-Leon M, Gomez-Polo M, Zeitler JM, Barmak AB, Kois JC, Perez-Barquero JA. Does the available interocclusal space influence the accuracy of the maxillomandibular relationship captured with an intraoral scanner? J Prosthet Dent. 2024 Aug;132(2):435-440. doi: 10.1016/j.prosdent.2022.09.004. Epub 2022 Oct 28. PMID 36349566
- [Background] Ries JM, Grunler C, Wichmann M, Matta RE. Three-dimensional analysis of the accuracy of conventional and completely digital interocclusal registration methods. J Prosthet Dent. 2022 Nov;128(5):994-1000. doi: 10.1016/j.prosdent.2021.03.005. Epub 2021 Apr 19. PMID 33888327
- [Background] Abdulateef S, Edher F, Hannam AG, Tobias DL, Wyatt CCL. Clinical accuracy and reproducibility of virtual interocclusal records. J Prosthet Dent. 2020 Dec;124(6):667-673. doi: 10.1016/j.prosdent.2019.11.014. Epub 2020 Feb 1. PMID 32014284
- [Background] Edher F, Hannam AG, Tobias DL, Wyatt CCL. The accuracy of virtual interocclusal registration during intraoral scanning. J Prosthet Dent. 2018 Dec;120(6):904-912. doi: 10.1016/j.prosdent.2018.01.024. Epub 2018 Jun 28. PMID 29961618
- [Background] Yee SHX, Esguerra RJ, Chew AAQ, Wong KM, Tan KBC. Three-Dimensional Static Articulation Accuracy of Virtual Models - Part I: System Trueness and Precision. J Prosthodont. 2018 Feb;27(2):129-136. doi: 10.1111/jopr.12723. Epub 2017 Dec 13. PMID 29235202
- [Background] Zimmermann M, Ender A, Attin T, Mehl A. Accuracy of Buccal Scan Procedures for the Registration of Habitual Intercuspation. Oper Dent. 2018 Nov/Dec;43(6):573-580. doi: 10.2341/17-272-C. Epub 2018 Apr 9. PMID 29630481
- [Background] Jaschouz S, Mehl A. Reproducibility of habitual intercuspation in vivo. J Dent. 2014 Feb;42(2):210-8. doi: 10.1016/j.jdent.2013.09.010. Epub 2013 Nov 2. PMID 24189225